CLINICAL TRIAL: NCT02366026
Title: REMUNE + AMPLIVAX IR103 HIV/AIDS Phase III Safety & Efficacy Study
Acronym: RAISE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Immune Response BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR103-007
Record Dates: First submitted 2015-02-06; First posted 2015-02-19 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: HIV
Keywords: HIV
MeSH Terms: interventions — IMO-2055; remune

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IR103 REMUNE + AMPLIVAX 1.0 (Experimental): IR103 Vaccine contain the same active component as REMUNE® (Inactivated HIV-1 Antigen Drug Substance at 10 μg/mL p24 dose), and have one dose of Amplivax™ (HYB2055) Adjuvant (1.0 mg) added before emulsification in Incomplete Freund's Adjuvant (the same adjuvant and in the same ratio that is used in REMUNE).
  Interventions: Biological: IR103
- AMPLIVAX 1.0 + IFA (Placebo Comparator): AMPLIVAX 1.0 mg Amplivax™ (HYB2055) Adjuvant (1.0 mg) + IFA Incomplete Freund's Adjuvant (the same adjuvant and in the same ratio that is used in REMUNE).
  Interventions: Biological: IR103

INTERVENTIONS:
Biological: IR103 — REMUNE HIV/AIDS Vaccine with two adjuvants IFA + Amplivax
  Other Names: HIV-1 IMMUNOGEN + Amplivax; REMUNE + Amplivax

SUMMARY:
The primary objective is to compare & evaluate between the treatment groups the changes in decline/reduction of HIV viral load changes in the Remune + Amplivax group vs the Amplivax placebo groups. Additional objectives include changes in WBC White Blood Cell counts & CD4+ & CD8+ T cell counts along with increased HIV immunity.

DETAILED DESCRIPTION:
This is a 500 subject Multi Center double-blind randomized, Safety & Efficacy, HIV/AIDS Phase III study, to primarily to evaluate the safety and efficacy of HIV-1 immunogen & Amplivax compared to placebo group Amplivax in viral load, and secondarily to examine changes in CD4+ & CD8+ T cell counts, determine Remune vaccines effect of multiple inoculations of HIV-1 immunogen + Amplivax on viral replication in adults with HIV-1 infection & to examine immunogenicity of Remune + Amplivax in a Multi-center, randomized , double-blind, placebo-controlled, two arm parallel design study of Remune + Amplivax.

ELIGIBILITY:
Inclusion Criteria:

* Are HIV-positive and started anti-HIV drugs soon after tests showed the presence of HIV.
* Are at least 16 years old (consent of parent or guardian required if under 18 years).

Exclusion Criteria:

* Healthy Subjects
* Currently abuse alcohol or drugs.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to compare & evaluate between the treatment groups the changes in HIV viral load at Week 52 | 52 Weeks
  The primary objective is to compare & evaluate between the treatment groups the changes in HIV viral load at Week 52

SECONDARY OUTCOMES:
The secondary objective is to evaluate & compare changes in WBC White Blood Cell counts between the treatment groups | 52 Weeks
  The secondary objective is to evaluate & compare changes in WBC White Blood Cell Counts between the treatment groups at Week 52
The secondary objective is to evaluate & compare changes in CD4+ & CD8+ T cell counts between the treatment groups | 52 Weeks
  The secondary objective is to evaluate & compare changes in CD4+ & CD8+ T cell counts between the treatment groups at Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bartholomew, PhD, Study Director — Immune Response BioPharma, Inc.
Locations (1):
- Clinical Site TBA, San Diego, California, United States